CLINICAL TRIAL: NCT01550757
Title: Aligning Resources to Care for Homeless Veterans (ARCH)
Brief Title: Aligning Resources to Care for Homeless Veterans
Acronym: ARCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SDR 11-230
Record Dates: First submitted 2011-09-13; First posted 2012-03-12 (Estimated); Results first posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-05

CONDITIONS: Homeless Persons; Primary Health Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (No Intervention): Normal PACT Clinical Care
- Arm 2 (Experimental): Normal PACT Clinical Care + Embedded Peer Mentor
  Interventions: Behavioral: Embedded Peer Mentor
- Arm 3 (No Intervention): Normal Homeless Oriented PACT Clinical Care
- Arm 4 (Experimental): Normal Homeless Oriented PACT Clinical Care + Embedded Peer Mentor
  Interventions: Behavioral: Embedded Peer Mentor

INTERVENTIONS:
Behavioral: Embedded Peer Mentor — This intervention/condition consists of a formerly homeless individual embedded in the PACT or H-PACT clinic team. This person is responsible for community-based follow-up for homeless patients randomly assigned to him or her. In addition to structured, scheduled meetings with assigned study subjects, the peer mentor will also participate in PACT/H-PACT team meetings and serve as a liaison between the study subject and his or her primary care team. Peer mentors will be hired as VA term employees in Research.
  Arms: Arm 2; Arm 4

SUMMARY:
"Aligning Resources to Care for Homeless Veterans" (ARCH) will study ways to best organize and deliver primary care for homeless Veterans. The investigators will assess 4 different adaptations of the PACT primary care model in a mixed methods study that includes multi-center, randomized-controlled trials of embedded peer-mentoring within different iterations of the PACT model, focus groups of study participants assessing satisfaction, treatment engagement and self-efficacy within the different care models and a cost-utility analysis to determine the most cost-efficient approach to organizing care for this population. Findings from this study will help determine optimal care approaches for reducing emergency department visits and acute hospitalizations, increasing patient satisfaction, and improving chronic disease management. Findings from this study will also substantively add to our understanding of health seeking behavior and the care of vulnerable/high-risk Veteran populations as well as clinical systems design. This project reflects a true "field-based study" to identify optimal and feasible approaches to patient care within our current VHA system. Finally, it will help inform pressing policy issues relevant to two identified T-21 priority areas: Ending Veteran Homelessness in 5 Years and Transforming to a Patient Centered Primary Care model.

DETAILED DESCRIPTION:
Background:

Primary care, and specifically primary care directed to homeless Veterans represents an opportunity to engage individuals in care, address unmet health needs and facilitate receipt of services necessary to exit homelessness. However, it is unclear what the best and most cost-efficient approach is to providing this care. Past research suggests two alternative approaches to organizing and delivering primary care to homeless Veterans: (1) structurally realigned and organized care and (2) embedded peer mentoring. The overall purpose of our research is to compare and contrast outcomes from 4 different adaptations and combinations of primary care delivery to homeless Veterans within the construct of the Patient Aligned Care Team (PACT) model for primary care.

Objectives:

1. To test whether a peer mentor intervention embedded in the Patient Aligned Care Team (PACT) model will be more effective than usual-care PACT or, in a separate randomized controlled trial, within a homeless-oriented PACT (H-PACT) model, in reducing emergency department use and hospitalizations, improving chronic disease management, and increasing participation in homeless programming.
2. To compare clinical outcomes, service use, treatment engagement, self-efficacy, and patient satisfaction of participants in usual care-PACT with and without peer mentoring to H-PACT with and without peer mentoring.
3. To determine differential costs and cost offsets associated with each PACT model adaptation in relation to care outcomes for homeless Veterans.
4. To determine whether a structurally adapted health care delivery model for homeless Veterans (homeless PACT) affects treatment engagement, as measured by utilization of services over time, compared with assignment to a general population Patient Aligned Care Team or no primary care assignment.

Methods:

Substudy #1- Two multi-center Randomized Controlled Trials: The first comparing PACT to PACT+Peer Support (PACT+P); and the second comparing Homeless-oriented PACT (H-PACT) to H-PACT+Peer Support (H-PACT+P). Within each site we will conduct a 1:1 RCT of embedded peer support.

Substudy #2- A qualitative study using focus groups of study participants from each of the intervention arms to assess perceptions of care, treatment engagement, and satisfaction within each approach. These findings will be triangulated with survey data and conditional logistic regression modeling to address the question of how each model is perceived by those receiving care within it and what outcomes can be ascribed to each care approach. This submission will occur at the end of Year 2 of the project and be specific for the focus group activities.

Substudy #3- Cost-Utilization Analysis Study: We will conduct a cost-utilization analysis assessing cost offsets using CPRS, DSS, and PCMM labor mapping data to develop cost models for each care approach.

Substudy #4- VINCI Data Extraction & Natural Language Processing: Use VINCI to analyze for PACT and H-PACT emergency department visits, including diagnosis, whether substance abuse was a factor, whether it resulted in a hospital admission, and what type of aftercare occurred (primary care follow-up, case manager telephone call note, etc.); hospital admissions (diagnosis, length of stay, and aftercare follow-up), ambulatory care utilization (primary care, mental health, specialty clinics, outpatient substance abuse treatment, and homeless programming - VRRC), including both face-to-face and remote-based care (My HealtheVet, telehealth, telephone notes), medication compliance with continuous prescriptions (i.e. insulin, antihypertensives), and chronic disease monitoring and management (blood pressure, diabetes care, hyperlipidemia in heart disease and diabetic patients). Baseline utilization (prior 6 months) of emergency department, inpatient and primary care prior to cohort tracking will be conducted to allow for post-hoc stratification of patient subgroups based on predicted risk for high use patterning.

ELIGIBILITY:
Inclusion Criteria:

* The study population will be homeless Veterans enrolled in primary care (including both new and established patients who are homeless at the time of enrollment).
* Currently homeless to include: unsheltered; staying in an emergency shelter; in transitional/Grant and Per Diem housing; or doubled-up with a family member or friend and not paying rent.

Exclusion Criteria:

* Currently enrolled in Mental Health Intensive Case Management (MHICM) or other VA-based case/care managed program;
* Stated plans to leave the area within 6 months of enrollment;
* Unable or unwilling to provide informed consent;
* Pregnant women will because excluded because we do not wish to detract from the amount of specialty care and services they receive and need.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P O'Toole, MD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

REFERENCES:
- [Background] Resnik L, Ekerholm S, Johnson EE, Ellison ML, O'Toole TP. Which Homeless Veterans Benefit From a Peer Mentor and How? J Clin Psychol. 2017 Sep;73(9):1027-1047. doi: 10.1002/jclp.22407. Epub 2016 Oct 20. PMID 27764527
- [Result] Yoon J, Lo J, Gehlert E, Johnson EE, O'Toole TP. Homeless Veterans' Use of Peer Mentors and Effects on Costs and Utilization in VA Clinics. Psychiatr Serv. 2017 Jun 1;68(6):628-631. doi: 10.1176/appi.ps.201600290. Epub 2017 Feb 1. PMID 28142391
- [Derived] Van Voorhees EE, Resnik L, Johnson E, O'Toole T. Posttraumatic stress disorder and interpersonal process in homeless veterans participating in a peer mentoring intervention: Associations with program benefit. Psychol Serv. 2019 Aug;16(3):463-474. doi: 10.1037/ser0000231. Epub 2018 Jan 25. PMID 29369660
- [Derived] Gundlapalli AV, Redd A, Bolton D, Vanneman ME, Carter ME, Johnson E, Samore MH, Fargo JD, O'Toole TP. Patient-aligned Care Team Engagement to Connect Veterans Experiencing Homelessness With Appropriate Health Care. Med Care. 2017 Sep;55 Suppl 9 Suppl 2:S104-S110. doi: 10.1097/MLR.0000000000000770. PMID 28806373

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Normal PACT Clinical Care: Normal Patient Aligned Care Team Clinical Care
- Arm 2: Normal PACT Clinical Care + Embedded Peer Mentor: Normal PACT Clinical Care + Embedded Peer Mentor
  Embedded Peer Mentor: This intervention/condition consists of a formerly homeless individual embedded in the PACT or H-PACT clinic team. This person is responsible for community-based follow-up for homeless patients randomly assigned to him or her. In addition to structured, scheduled meetings with assigned study subjects, the peer mentor will also participate in PACT/H-PACT team meetings and serve as a liaison between the study subject and his or her primary care team. Peer mentors will be hired as VA term employees in Research.
- Arm 3: Normal Homeless Oriented PACT Clinical Care: Normal Homeless Oriented Patient Aligned Care Team Clinical Care
- Arm 4: Normal Homeless Oriented PACT Clinical Care + Embedded: Normal Homeless Oriented PACT Clinical Care + Embedded Peer Mentor
  Embedded Peer Mentor: This intervention/condition consists of a formerly homeless individual embedded in the PACT or H-PACT clinic team. This person is responsible for community-based follow-up for homeless patients randomly assigned to him or her. In addition to structured, scheduled meetings with assigned study subjects, the peer mentor will also participate in PACT/H-PACT team meetings and serve as a liaison between the study subject and his or her primary care team. Peer mentors will be hired as VA term employees in Research.
Period: Overall Study
Arm/Group | Arm 1: Normal PACT Clinical Care | Arm 2: Normal PACT Clinical Care + Embedded Peer Mentor | Arm 3: Normal Homeless Oriented PACT Clinical Care | Arm 4: Normal Homeless Oriented PACT Clinical Care + Embedded
Started | 56 | 52 | 130 | 144
Completed | 33 | 38 | 85 | 90
Not Completed | 23 | 14 | 45 | 54
Not completed — Lost to Follow-up | 21 | 14 | 42 | 53
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Normal PACT Clinical Care | Arm 2: Normal PACT Clinical Care + Embedded Peer Mentor | Arm 3: Normal Homeless Oriented PACT Clinical Care | Arm 4: Normal Homeless Oriented PACT Clinical Care + Embedded | Total
Number analyzed (Participants) | 56 | 52 | 130 | 144 | 382
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 49 | 120 | 130 | 351
  >=65 years | 4 | 3 | 10 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (8.8) | 50.3 (10.0) | 51.2 (9.5) | 52.6 (9.4) | 52.2 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 2 | 6 | 16
  Male | 49 | 51 | 128 | 138 | 366
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 128 | 138 | 366

OUTCOME MEASURES:

1. Primary Outcome: A Primary Outcome for This Study is the Number of Non-acute Emergency Department Visits.
Description: A primary outcome for this study is non-acute emergency department visits.
Time Frame: Two years.
Population: Veterans enrolled in the study based on the type of care they received at VA and then randomized to receive a peer or not.
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Arm 1: Normal PACT Clinical Care | Arm 2: Normal PACT Clinical Care + Embedded Peer Mentor | Arm 3: Normal Homeless Oriented PACT Clinical Care | Arm 4: Normal Homeless Oriented PACT Clinical Care + Embedded
Number analyzed (Participants) | 56 | 52 | 130 | 144
number of visits | 1.1 (1.6) | 0.8 (2.3) | 0.7 (1.2) | 1.0 (1.7)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during active enrollment in the randomized controlled trial, May 2012 - March 2014 (22 months).
Description: We submitted an amendment about adverse events. It outlined "expected AEs" commonly seen in the homeless population. As this study is considered "low risk" and unrelated to specific disease management, we defined the medical management issues/expected hospitalizations we anticipated among our homeless cohort. In accordance with all VA policies, we report all unexpected events occurring during study participation, events impacting research staff, and any events involving research privacy.
Arm/Group | Arm 1: Normal PACT Clinical Care | Arm 2: Normal PACT Clinical Care + Embedded Peer Mentor | Arm 3: Normal Homeless Oriented PACT Clinical Care | Arm 4: Normal Homeless Oriented PACT Clinical Care + Embedded
All-Cause Mortality (participants affected / at risk) | 1/56 | 0/52 | 1/130 | 1/144
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/52 | 0/130 | 0/144
Other Adverse Events (participants affected / at risk) | 0/56 | 0/52 | 0/130 | 0/144

LIMITATIONS AND CAVEATS:
All AE and SAE monitoring was discussed with and approved by all regulatory authorities (IRB, DSMB, and research compliance officer).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes